CLINICAL TRIAL: NCT00558259
Title: Twice-daily Oral Direct Thrombin Inhibitor Dabigatran Etexilate in the Long-term Prevention of Recurrent Symptomatic Proximal Venous Thromboembolism in Patients With Symptomatic Deep-vein Thrombosis or Pulmonary Embolism.
Brief Title: Twice-daily Oral Direct Thrombin Inhibitor Dabigatran Etexilate in the Long Term Prevention of Recurrent Symptomatic VTE
Acronym: RE-SONATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1160.63; 2007-002586-12 (EudraCT Number: EudraCT)
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Results first posted 2012-03-02 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-02

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Dabigatran

ARMS (2):
- dabigatran etexilate 150 mg BID (Experimental): Patient to receive dabigatran etexilatate capsules 150 mg twice daily
  Interventions: Drug: dabigatran etexilate 150 mg twice daily (BID)
- matching placebo twice daily (BID) (Placebo Comparator): Patient to receive dabigatran extexilate matching placebo capsules twice daily
  Interventions: Drug: matching placebo twice daily (BID)

INTERVENTIONS:
Drug: dabigatran etexilate 150 mg twice daily (BID) — dabigatran etexilate capsules 150 mg BID
  Arms: dabigatran etexilate 150 mg BID
Drug: matching placebo twice daily (BID) — Matching placebo BID
  Arms: matching placebo twice daily (BID)

SUMMARY:
The primary efficacy objective is to evaluate whether dabigatran etexilate is superior to placebo in the long-term prevention of recurrent symptomatic venous thrombo-embolism (VTE) in patients with symptomatic deep-vein thrombosis (DVT) or pulmonary embolism (PE) who completed 6 to 18 months of treatment with vitamin K antagonist (VKA).

ELIGIBILITY:
Inclusion criteria:

1. Patients with confirmed symptomatic PE or proximal DVT of the leg(s) who have been treated for 6 to 18 months with therapeutic dosages (intended INR between 2-3) of an oral VKA (e.g. warfarin, acenocoumarol, phenprocoumon, or fluindione) or RE-COVER study medication up to the moment of screening for the current study.
2. Written informed consent

Exclusion criteria:

1. Younger then 18 years of age
2. Indication for VKA other than DVT and/or PE
3. Patients in whom anticoagulant treatment for their index PE or DVT should be continued
4. Active liver disease or liver disease decreasing survival (e.g. acute hepatitis, chronic active hepatitis, cirrhosis) or ALAT > 3 x ULN
5. Creatinine clearance < 30 ml/min
6. Acute bacterial endocarditis
7. Active bleeding or high risk for bleeding.
8. Uncontrolled hypertension (investigators judgement)
9. Intake of another experimental drug within the 30 days prior to randomization into the study
10. Life expectancy <6 months
11. Childbearing potential without proper contraceptive measures*, pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1353 (Actual)
Dates: Start 2007-11; Primary Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (147):
- United States (21):
  - 1160.63.01025 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1160.63.01023 Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - 1160.63.01002 Boehringer Ingelheim Investigational Site, Laguna Hills, California
  - 1160.63.01014 Boehringer Ingelheim Investigational Site, Colorado Springs, Colorado
  - 1160.63.01003 Boehringer Ingelheim Investigational Site, Jacksonville, Florida
  - 1160.63.01030 Boehringer Ingelheim Investigational Site, Key West, Florida
  - 1160.63.01022 Boehringer Ingelheim Investigational Site, Lafayette, Louisiana
  - 1160.63.01044 Boehringer Ingelheim Investigational Site, New Iberia, Louisiana
  - 1160.63.01017 Boehringer Ingelheim Investigational Site, Biddeford, Maine
  - 1160.63.01004 Boehringer Ingelheim Investigational Site, Salisbury, Maryland
  - 1160.63.01016 Boehringer Ingelheim Investigational Site, Worcester, Massachusetts
  - 1160.63.01037 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1160.63.01019 Boehringer Ingelheim Investigational Site, Missoula, Montana
  - 1160.63.01032 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1160.63.01001 Boehringer Ingelheim Investigational Site, Uniontown, Pennsylvania
  - 1160.63.01024 Boehringer Ingelheim Investigational Site, Uniontown, Pennsylvania
  - 1160.63.01005 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1160.63.01020 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1160.63.01011 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 1160.63.01007 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1160.63.01035 Boehringer Ingelheim Investigational Site, Bellevue, Washington
- Australia (4):
  - 1160.63.61002 Boehringer Ingelheim Investigational Site, Greenslopes, Queensland
  - 1160.63.61003 Boehringer Ingelheim Investigational Site, Elizabeth Vale, South Australia
  - 1160.63.61001 Boehringer Ingelheim Investigational Site, Clayton, Victoria
  - 1160.63.61004 Boehringer Ingelheim Investigational Site, Nedlands, Western Australia
- Austria (5):
  - 1160.63.43005 Boehringer Ingelheim Investigational Site, Graz
  - 1160.63.43006 Boehringer Ingelheim Investigational Site, Innsbruck
  - 1160.63.43001 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.63.43002 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.63.43004 Boehringer Ingelheim Investigational Site, Vienna
- Belgium (5):
  - 1160.63.32005 Boehringer Ingelheim Investigational Site, Aalst
  - 1160.63.32004 Boehringer Ingelheim Investigational Site, Duffel
  - 1160.63.32003 Boehringer Ingelheim Investigational Site, Kortrijk
  - 1160.63.32001 Boehringer Ingelheim Investigational Site, Leuven
  - 1160.63.32002 Boehringer Ingelheim Investigational Site, Lier
- Canada (4):
  - 1160.63.02013 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1160.63.02004 Boehringer Ingelheim Investigational Site, Saint John, New Brunswick
  - 1160.63.02005 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1160.63.02020 Boehringer Ingelheim Investigational Site, Québec, Quebec
- Czechia (14):
  - 1160.63.42004 Boehringer Ingelheim Investigational Site, České Budějovice
  - 1160.63.42003 Boehringer Ingelheim Investigational Site, Jablonec nad Nisou
  - 1160.63.42008 Boehringer Ingelheim Investigational Site, Kladno
  - 1160.63.42012 Boehringer Ingelheim Investigational Site, Liberec
  - 1160.63.42010 Boehringer Ingelheim Investigational Site, Nymburk
  - 1160.63.42009 Boehringer Ingelheim Investigational Site, Ostrava
  - 1160.63.42011 Boehringer Ingelheim Investigational Site, Ostrava-Vitkovice
  - 1160.63.42001 Boehringer Ingelheim Investigational Site, Prague
  - 1160.63.42006 Boehringer Ingelheim Investigational Site, Prague
  - 1160.63.42002 Boehringer Ingelheim Investigational Site, Prague 4-Krc
  - 1160.63.42005 Boehringer Ingelheim Investigational Site, Prostějov
  - 1160.63.42007 Boehringer Ingelheim Investigational Site, Rakovník
  - 1160.63.42013 Boehringer Ingelheim Investigational Site, Slaný
  - 1160.63.42014 Boehringer Ingelheim Investigational Site, Tábor
- Estonia (3):
  - 1160.63.37202 Boehringer Ingelheim Investigational Site, Kohtla-Järve
  - 1160.63.37203 Boehringer Ingelheim Investigational Site, Tallinn
  - 1160.63.37201 Boehringer Ingelheim Investigational Site, Tartu
- Germany (9):
  - 1160.63.49013 Boehringer Ingelheim Investigational Site, Darmstadt
  - 1160.63.49017 Boehringer Ingelheim Investigational Site, Dresden
  - 1160.63.49018 Boehringer Ingelheim Investigational Site, Dresden
  - 1160.63.49014 Boehringer Ingelheim Investigational Site, Giessen
  - 1160.63.49011 Boehringer Ingelheim Investigational Site, Ludwigshafen
  - 1160.63.49005 Boehringer Ingelheim Investigational Site, Mannheim
  - 1160.63.49010 Boehringer Ingelheim Investigational Site, Mannheim
  - 1160.63.49007 Boehringer Ingelheim Investigational Site, München
  - 1160.63.49009 Boehringer Ingelheim Investigational Site, Püttlingen
- Italy (18):
  - 1160.63.39006 Boehringer Ingelheim Investigational Site, Bergamo
  - 1160.63.39015 Boehringer Ingelheim Investigational Site, Castelfranco Veneto (TV)
  - 1160.63.39019 Boehringer Ingelheim Investigational Site, Chieti Scalo (CH)
  - 1160.63.39003 Boehringer Ingelheim Investigational Site, Cosenza
  - 1160.63.39008 Boehringer Ingelheim Investigational Site, Fidenza (PR)
  - 1160.63.39011 Boehringer Ingelheim Investigational Site, Florence
  - 1160.63.39009 Boehringer Ingelheim Investigational Site, Genova
  - 1160.63.39004 Boehringer Ingelheim Investigational Site, Milan
  - 1160.63.39010 Boehringer Ingelheim Investigational Site, Milan
  - 1160.63.39020 Boehringer Ingelheim Investigational Site, Milan
  - 1160.63.39022 Boehringer Ingelheim Investigational Site, Napoli
  - 1160.63.39001 Boehringer Ingelheim Investigational Site, Palermo
  - 1160.63.39007 Boehringer Ingelheim Investigational Site, Pisa
  - 1160.63.39012 Boehringer Ingelheim Investigational Site, Rimini
  - 1160.63.39017 Boehringer Ingelheim Investigational Site, Roma
  - 1160.63.39014 Boehringer Ingelheim Investigational Site, Treviso
  - 1160.63.39002 Boehringer Ingelheim Investigational Site, Udine
  - 1160.63.39016 Boehringer Ingelheim Investigational Site, Vittorio Veneto (TV)
- Latvia (2):
  - 1160.63.37101 Boehringer Ingelheim Investigational Site, Daugavpils
  - 1160.63.37102 Boehringer Ingelheim Investigational Site, Riga
- Lithuania (2):
  - 1160.63.37002 Boehringer Ingelheim Investigational Site, Kaunas
  - 1160.63.37001 Boehringer Ingelheim Investigational Site, Vilnius
- Netherlands (9):
  - 1160.63.31010 Boehringer Ingelheim Investigational Site, Assen
  - 1160.63.31006 Boehringer Ingelheim Investigational Site, Breda
  - 1160.63.31011 Boehringer Ingelheim Investigational Site, Den Helder
  - 1160.63.31012 Boehringer Ingelheim Investigational Site, Dirksland
  - 1160.63.31003 Boehringer Ingelheim Investigational Site, Eindhoven
  - 1160.63.31001 Boehringer Ingelheim Investigational Site, Groningen
  - 1160.63.31009 Boehringer Ingelheim Investigational Site, Heerlen
  - 1160.63.31008 Boehringer Ingelheim Investigational Site, Oss
  - 1160.63.31007 Boehringer Ingelheim Investigational Site, The Hague
- 1160.63.64002 Boehringer Ingelheim Investigational Site, Christchurch, New Zealand
- Poland (9):
  - 1160.63.48010 Boehringer Ingelheim Investigational Site, Kielce
  - 1160.63.48003 Boehringer Ingelheim Investigational Site, Poznan
  - 1160.63.48001 Boehringer Ingelheim Investigational Site, Warsaw
  - 1160.63.48002 Boehringer Ingelheim Investigational Site, Warsaw
  - 1160.63.48004 Boehringer Ingelheim Investigational Site, Warsaw
  - 1160.63.48005 Boehringer Ingelheim Investigational Site, Warsaw
  - 1160.63.48006 Boehringer Ingelheim Investigational Site, Warsaw
  - 1160.63.48007 Boehringer Ingelheim Investigational Site, Warsaw
  - 1160.63.48008 Boehringer Ingelheim Investigational Site, Warsaw
- Russia (5):
  - 1160.63.07004 Boehringer Ingelheim Investigational Site, Kursk
  - 1160.63.07014 Boehringer Ingelheim Investigational Site, Ufa
  - 1160.63.07005 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 1160.63.07006 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 1160.63.07007 Boehringer Ingelheim Investigational Site, Yekaterinburg
- 1160.63.65001 Boehringer Ingelheim Investigational Site, Singapore, Singapore
- South Africa (4):
  - 1160.63.27003 Boehringer Ingelheim Investigational Site, Cape Town
  - 1160.63.27007 Boehringer Ingelheim Investigational Site, Centurion
  - 1160.63.27009 Boehringer Ingelheim Investigational Site, Krugersdorp
  - 1160.63.27001 Boehringer Ingelheim Investigational Site, Somerset West
- South Korea (9):
  - 1160.63.82010 Boehringer Ingelheim Investigational Site, Gwangju
  - 1160.63.82003 Boehringer Ingelheim Investigational Site, Incheon
  - 1160.63.82005 Boehringer Ingelheim Investigational Site, Kyeonggi-do
  - 1160.63.82001 Boehringer Ingelheim Investigational Site, Kyunggi-do
  - 1160.63.82004 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.63.82006 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.63.82008 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.63.82011 Boehringer Ingelheim Investigational Site, Seoul
  - 1160.63.82007 Boehringer Ingelheim Investigational Site, Suwon
- Sweden (7):
  - 1160.63.46001 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1160.63.46006 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1160.63.46002 Boehringer Ingelheim Investigational Site, Lund
  - 1160.63.46004 Boehringer Ingelheim Investigational Site, Mölndal
  - 1160.63.46007 Boehringer Ingelheim Investigational Site, Skövde
  - 1160.63.46005 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.63.46003 Boehringer Ingelheim Investigational Site, Värnamo
- Switzerland (11):
  - 1160.63.41012 Boehringer Ingelheim Investigational Site, Basel
  - 1160.63.41011 Boehringer Ingelheim Investigational Site, Bruderholz
  - 1160.63.41003 Boehringer Ingelheim Investigational Site, Cham
  - 1160.63.41001 Boehringer Ingelheim Investigational Site, Glarus
  - 1160.63.41014 Boehringer Ingelheim Investigational Site, Lucerne
  - 1160.63.41016 Boehringer Ingelheim Investigational Site, Lucerne
  - 1160.63.41005 Boehringer Ingelheim Investigational Site, Schiers
  - 1160.63.41009 Boehringer Ingelheim Investigational Site, Thun
  - 1160.63.41022 Boehringer Ingelheim Investigational Site, Wetzikon
  - 1160.63.41008 Boehringer Ingelheim Investigational Site, Zug
  - 1160.63.41006 Boehringer Ingelheim Investigational Site, Zurich
- Thailand (4):
  - 1160.63.66002 Boehringer Ingelheim Investigational Site, Bangkok
  - 1160.63.66003 Boehringer Ingelheim Investigational Site, Bangkok
  - 1160.63.66004 Boehringer Ingelheim Investigational Site, Bangkok
  - 1160.63.66001 Boehringer Ingelheim Investigational Site, Chiang Mai

REFERENCES:
- [Derived] Majeed A, Hwang HG, Connolly SJ, Eikelboom JW, Ezekowitz MD, Wallentin L, Brueckmann M, Fraessdorf M, Yusuf S, Schulman S. Management and outcomes of major bleeding during treatment with dabigatran or warfarin. Circulation. 2013 Nov 19;128(21):2325-32. doi: 10.1161/CIRCULATIONAHA.113.002332. Epub 2013 Sep 30. PMID 24081972
- [Derived] Schulman S, Kearon C, Kakkar AK, Schellong S, Eriksson H, Baanstra D, Kvamme AM, Friedman J, Mismetti P, Goldhaber SZ; RE-MEDY Trial Investigators; RE-SONATE Trial Investigators. Extended use of dabigatran, warfarin, or placebo in venous thromboembolism. N Engl J Med. 2013 Feb 21;368(8):709-18. doi: 10.1056/NEJMoa1113697. PMID 23425163

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 3 patients randomised to placebo who received Dabigatran only. For all analyses of efficacy, these patients are analysed as randomised. For all analyses of safety, these patients are analysed as treated.
Groups:
- Dabigatran: Dabigatran 150mg bid (twice daily)
- Placebo: Matching placebo
Period: Overall Study
Arm/Group | Dabigatran | Placebo
Started | 681 (Number who started treatment. There were 4 patients randomised to Dabigatran and not treated.) | 662 (Number who started treatment. There were 6 patients randomised to placebo and not treated.)
Completed | 610 (Completed treatment.) | 563 (Completed treatment.)
Not Completed | 71 | 99
Not completed — Adverse Event | 50 | 81
Not completed — Protocol Violation | 9 | 5
Not completed — Withdrawal by Subject | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Dabigatran: Dabigatran 150mg bid
- Total: Total of all reporting groups
Arm/Group | Dabigatran | Placebo | Total
Number analyzed (Participants) | 681 | 662 | 1343
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.1 (15.5) | 55.5 (15.1) | 55.8 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 300 | 298 | 598
  Male | 381 | 364 | 745
Body mass index (BMI) continuous [Mean (Standard Deviation); unit: kg/m^2] | 28.45 (5.44) | 28.41 (5.56) | 28.43 (5.50)

OUTCOME MEASURES:

1. Primary Outcome: Centrally Confirmed Symptomatic Recurrent Venous Thrombotic Events (VTE) Including Unexplained Death During the Intended Treatment Period
Description: Symptomatic recurrent VTE is the composite of recurrent deep vein thrombosis (DVT) , fatal or non-fatal pulmonary embolism (PE). Whilst the endpoint is time to event, the measured values present the number of participant with event and the hazard ratio presents the time to event.
Time Frame: 6 months
Population: Full analysis set (FAS) and analysed as randomised. FAS is defined as randomised and treated.
Measure: Number; unit: Participants
Arm/Group | Dabigatran | Placebo
Number analyzed (Participants) | 681 | 662
Participants | 3 (0.0) | 37 (0.0)
Statistical Analysis 1: Comparison: Dabigatran vs Placebo; Dabigatran vs placebo; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.08, 95% CI [0.02 to 0.25], Standard Error of Mean 0.05

2. Secondary Outcome: Centrally Confirmed Symptomatic Recurrent Venous Thrombotic Events (VTE) Excluding Unexplained Death During the Intended Treatment Period
Description: as for outcome 1
Time Frame: 6 months
Population: FAS and analysed as randomised.
Measure: Number; unit: Participants
Arm/Group | Dabigatran | Placebo
Number analyzed (Participants) | 681 | 662
Participants | 3 | 35
Statistical Analysis 1: Comparison: Dabigatran vs Placebo; Dabigatran vs placebo; Test type: Superiority or Other; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.08, 95% CI [0.03 to 0.27], Standard Error of Mean 0.05

3. Secondary Outcome: Centrally Confirmed Symptomatic Recurrent Deep Venous Thrombotic (DVT) Events During the Intended Treatment Period
Description: Number of the participants with centrally confirmed symptomatic recurrent deep venous thrombotic (DVT) events during the intended treatment period were described.
Time Frame: 6 months
Population: FAS and analysed as randomised.
Measure: Number; unit: Participants
Arm/Group | Dabigatran | Placebo
Number analyzed (Participants) | 681 | 662
Participants | 2 | 23
Statistical Analysis 1: Comparison: Dabigatran vs Placebo; Test type: Superiority or Other; p < 0.0001, Fisher Exact
Statistical Analysis 2: Comparison: Dabigatran; Test type: Superiority or Other; Percentage of participants with events = 0.3, 95% CI 2-sided [0.04 to 1.06] — The confidence interval (Clopper-Pearson method) was calculated for the percentage of participants experiencing DVT in Dabigatran group
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority or Other; Percentage of participants with events = 3.5, 95% CI 2-sided [2.21 to 5.17] — The confidence interval (Clopper-Pearson method) was calculated for the percentage of participants experiencing DVT in placebo group

4. Secondary Outcome: Centrally Confirmed Symptomatic Pulmonary Embolism (PE) Events During the Intended Treatment Period
Description: Number of participants with centrally confirmed symptomatic pulmonary embolism (PE) events during the intended treatment period were described.
Time Frame: 6 months
Population: FAS and analysed as randomised.
Measure: Number; unit: Participants
Arm/Group | Dabigatran | Placebo
Number analyzed (Participants) | 681 | 662
Participants | 1 | 14
Statistical Analysis 1: Comparison: Dabigatran vs Placebo; Dabigatran vs. Placebo; Test type: Superiority or Other; p = 0.0004, Fisher Exact
Statistical Analysis 2: Comparison: Dabigatran; Test type: Superiority or Other; Percentage of participants with events = 0.1, 95% CI 2-sided [0.00 to 0.82] — The confidence interval (Clopper-Pearson method) was calculated for the percentage of participants experiencing PE in Dabigatran group
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority or Other; Percentage of participants with events = 2.1, 95% CI 2-sided [1.16 to 3.52] — The confidence interval (Clopper-Pearson method) was calculated for the percentage of participants experiencing PE in placebo group

5. Secondary Outcome: Centrally Confirmed Unexplained Deaths During the Intended Treatment Period
Description: Number of participants with centrally confirmed unexplained deaths during the intended treatment period were described.
Time Frame: 6 months
Population: FAS and analysed as randomised.
Measure: Number; unit: participants
Arm/Group | Dabigatran | Placebo
Number analyzed (Participants) | 681 | 662
participants | 0 | 2
Statistical Analysis 1: Comparison: Dabigatran vs Placebo; Dabigatran vs. Placebo; Test type: Superiority or Other; p = 0.2428, Fisher Exact
Statistical Analysis 2: Comparison: Dabigatran; Test type: Superiority or Other; Percentage of participants with events = 0.0, 95% CI 2-sided [0.00 to 0.54] — The confidence interval (Clopper-Pearson method) was calculated for the percentage of participants with unexplained death in Dabigatran group
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority or Other; Percentage of participants with events = 0.3, 95% CI 2-sided [0.04 to 1.09] — The confidence interval (Clopper-Pearson method) was calculated for the percentage of participants with unexplained death in placebo group

6. Secondary Outcome: Centrally Confirmed Bleeding Event During the Treatment Period
Description: Major bleeding events (MBE) had to fulfil at least 1 of the following criteria:
  * Fatal bleeding
  * Associated with a fall in haemoglobin of ≥2 g/dL
  * Led to the transfusion of ≥2 units packed cells or whole blood
  * Occurred in a critical site: intracranial, intraspinal, intraocular, pericardial, intra-articular, intramuscular with compartment syndrome, retroperitoneal
  Other clinically relevant bleeding was defined as overt bleeding not meeting the criteria for an MBE but associated with medical intervention, unscheduled contact with a physician, (temporary) cessation of study treatment, or associated with discomfort such as pain, or impairment of activities of daily life.
  Examples of these bleedings were:
  * Bleeding that compromised haemodynamics
  * Bleeding that led to hospitalisation
  Trivial bleeding events were defined as all other bleeding events that did not fulfil the criteria of MBEs or CRBEs.
  All bleeding events include MBEs, CRBEs, and trivial bleeding events.
Time Frame: 6 months
Population: FAS and analysed as treated. There were 3 participants who were randomised to placebo but treated with dabigatran only.
Measure: Number; unit: participants
Arm/Group | Dabigatran | Placebo
Number analyzed (Participants) | 684 | 659
participants
  MBE | 2 | 0
  MBE or CRBE | 36 | 12
  All Bleeding | 72 | 39
Statistical Analysis 1: Comparison: Dabigatran vs Placebo; Dabigatran vs. Placebo - Analysis of time to first occurrence of an MBE during the treatment period - FAS - as treated; Test type: Superiority or Other; p = 0.4998, Fisher Exact — As the Cox model did not converge due to too few events, hazard ratios are not estimable
Statistical Analysis 2: Comparison: Dabigatran; Test type: Superiority or Other; Percentage of participants with events = 0.3, 95% CI 2-sided [0.04 to 1.05] — The confidence interval (Clopper-Pearson method) was calculated for the percentage of participants experiencing MBE in Dabigatran group
Statistical Analysis 3: Comparison: Placebo; Test type: Superiority or Other; Percentage of participants with events = 0.0, 95% CI 2-sided [0.00 to 0.56] — The confidence interval (Clopper-Pearson method) was calculated for the percentage of participants experiencing MBE in placebo group
Statistical Analysis 4: Comparison: Dabigatran vs Placebo; Dabigatran vs. Placebo- Analysis of time to first occurrence of a MBE or CRBE during the treatment period - FAS - as treated; Test type: Superiority or Other; p = 0.0013, Regression, Cox; Hazard Ratio (HR) = 2.92, 95% CI 2-sided [1.52 to 5.60], Standard Error of Mean 0.97
Statistical Analysis 5: Comparison: Dabigatran vs Placebo; Dabigatran vs. Placebo- Analysis of time to first occurrence of any bleeding event during the treatment period - FAS - as treated; Test type: Superiority or Other; p = 0.0027, Regression, Cox; Hazard Ratio (HR) = 1.82, 95% CI 2-sided [1.23 to 2.68], Standard Error of Mean 0.36

7. Secondary Outcome: Centrally Confirmed Cardiovascular Events During the Treatment Period
Description: Cardiovascular events that occurred during the treatment period + 3 days were summarised by treatment groups.
Time Frame: 6 months
Population: FAS and analysed as treated. There were 3 participants who were randomised to placebo but treated with dabigatran only.
Measure: Number; unit: participants
Arm/Group | Dabigatran | Placebo
Number analyzed (Participants) | 684 | 659
participants | 3 | 2

8. Secondary Outcome: Laboratory Measures, Especially Liver Function Tests (LFTs)
Description: Number of participants with possible clinically significant abnormalities during the treatment period.
Time Frame: 6 months
Population: FAS - As Treated Assignment
Measure: Number; unit: participants
Arm/Group | Dabigatran | Placebo
Number analyzed (Participants) | 684 | 659
participants
  AST increase (N=655, 629) | 2 | 2
  ALT increase (N=655, 629) | 3 | 5
  Alkaline phosphatase increase (N=658, 629) | 0 | 0
  Total bilirubin increase (N=658, 628) | 1 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Description: There were 3 patients who were randomised to placebo but who were treated with dabigatran only.
Arm/Group | Dabigatran | Placebo
Serious Adverse Events (participants affected / at risk) | 47/684 | 60/659
Other Adverse Events (participants affected / at risk) | 0/684 | 0/659
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran (N=684) | Placebo (N=659)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Amaurosis fugax (Eye disorders) | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 2 | 1
Oedema (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Polyp (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Unevaluable event (General disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2
Salmonella bacteraemia (Infections and infestations) | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 3
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 | 0
Diabetic hyperglycaemic coma (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 1 | 0
Personality disorder (Psychiatric disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 16
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Abdominal wall operation (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 15
Embolism venous (Vascular disorders) | 0 | 1
Essential hypertension (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.